CLINICAL TRIAL: NCT05461872
Title: Retrospective Review on PAEDIATRIC and ADOLESCENT ADNEXAL MASSES
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, NG Karen, Assistant Professor, Chinese University of Hong Kong
Other Study IDs: CRE 2022.205
Record Dates: First submitted 2022-06-23; First posted 2022-07-18 (Actual); Last update posted 2022-08-15 (Actual); Status verified 2022-08

CONDITIONS: Adnexal Mass
Keywords: Paediatric; ovarian cyst; ovarian tumor; torsion; adolescent adnexal mass
MeSH Terms: conditions — Ovarian Cysts; Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- girls with adnexal mass: All girls who presented with adnexal mass from 0-21 years old (inclusive).
  Subjects will be identified from review of clinical records.
  Girl aged 21 or below who attended the NTEC cluster from 1990-2021 with available medical records.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
To review the characteristic, presentation and outcome of girls presented with adnexal masses to hopefully develop a management algorithm for girls with adnexal masses.

DETAILED DESCRIPTION:
Background, current evidence and key references:

In paediatric and adolescent girls, preservation of the ovaries for those suffering from ovarian masses requiring surgery is important to maximize future fertility. However, when one faces an ovarian mass in a girl, on one hand, there is potential fertility compromise in those who had extensive ovarian surgery, on the other hand there is a small but non-negligible potential malignancy risk. There are distinct differences in pathologies and imaging findings in girls compared to adults. There arises the question on the most suitable way to triage children for the suitable management, be it conservative, ovarian preserving or more radical surgery.

There have been different diagnostic tools developed to aid the evaluation of adnexal masses in women with only limited evidence on the usage of these tools when being applied to the paediatric and adolescent age group. Attempts have been made in creating treatment guidelines for children, however no prospective randomized trials exist in this area. Therefore, it is important to identify and develop the most suitable triage algorithm for this group of patients.

Aim of study:

In this study, we aim to review the presentation, participant characteristics, imaging findings and histopathological findings, and validate the applicability of the various diagnostic tools in the paediatric and adolescent population to hopefully develop a management algorithm to improve the ovarian preservation rate without jeopardizing the potential malignancy risk in girls with adnexal masses.

Aim to look at whether adult scoring systems for adnexal mass can be applied to the paediatric and adolescent population to differentiate between benign and malignant adnexal masses.

Hypothesis:

The current diagnostic algorithms available for adults are applicable to the paediatric and adolescent population.

Outcome measure:

Participant characteristics, imaging findings, biochemical markers, operative record and histopathological findings, post-operative complications, post-operative menstrual symptoms, and any subsequent reproductive outcome.

Methods of Data Analysis:

The presentation, characteristics, imaging prior to surgery, surgical approaches, histopathological diagnosis and outcome of participant who presented with adnexal masses will be reviewed. The findings according to the data obtained from the review of medical records will be compared to the pre-existing rules and management algorithm for adults. The scoring systems or algorithms will then be validated with histopathological findings or participant outcome to assess applicability in our study population.

SPSS statistical program (SPSS Inc. version 21; IBM Corp., Armonk, NY, USA) was used to analyse the data collected. Normally distributed data was described using means (SD), whereas non-normally distributed data were described using medians (range).

A probability value of <0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* girls who presented with adnexal mass
* aged 0-21 years old

Exclusion Criteria:

* Girls older than 21 years old

Ages: 1 Day to 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — All girls who presented with adnexal mass from 0-21 years old (inclusive)
Study Population: Expecting number of record will be reviewed: 300.
  Participant will be identified from review of clinical records.
  Participants aged 21 or below who attended the NTEC cluster from 1990-2021 with available medical records.
  Since not all data are available in each case, expecting 300 patient records will be reviewed to have target 139 completed record.
  Total number of females from HK census in 2021: 0-19 years old: 521857 9-11% are malignant
  Sample size calculation work with a 95% confidence level; Confidence interval (margin of error) of ± 5%; Population portion of 10% Population size: 521857
  Sample size=139
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-08-12 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
To review the characteristic of girls presented with adnexal masses to hopefully develop a management algorithm for girls with adnexal masses. | Baseline
  To review the characteristic of girls presented with adnexal masses to hopefully develop a management algorithm for girls with adnexal masses.
To review the imaging findings of girls presented with adnexal masses to hopefully develop a management algorithm for girls with adnexal masses. | Baseline
  To review the imaging findings of girls presented with adnexal masses to hopefully develop a management algorithm for girls with adnexal masses.
To review the biochemical markers of girls presented with adnexal masses to hopefully develop a management algorithm for girls with adnexal masses. | Baseline
  To review the biochemical markers of girls presented with adnexal masses to hopefully develop a management algorithm for girls with adnexal masses.
To review the operative record of girls presented with adnexal masses to hopefully develop a management algorithm for girls with adnexal masses. | Baseline
  To review the operative record of girls presented with adnexal masses to hopefully develop a management algorithm for girls with adnexal masses.
To review the histopathological findings of girls presented with adnexal masses to hopefully develop a management algorithm for girls with adnexal masses. | Baseline
  To review the histopathological findings of girls presented with adnexal masses to hopefully develop a management algorithm for girls with adnexal masses.
To review the post-operative complications of girls presented with adnexal masses to hopefully develop a management algorithm for girls with adnexal masses. | Baseline
  To review the post-operative complications of girls presented with adnexal masses to hopefully develop a management algorithm for girls with adnexal masses.
To review the post-operative menstrual symptoms of girls presented with adnexal masses to hopefully develop a management algorithm for girls with adnexal masses. | Baseline
  To review the post-operative menstrual symptoms of girls presented with adnexal masses to hopefully develop a management algorithm for girls with adnexal masses.
To review the subsequent reproductive outcome of girls presented with adnexal masses to hopefully develop a management algorithm for girls with adnexal masses. | Baseline
  To review the subsequent reproductive outcome of girls presented with adnexal masses to hopefully develop a management algorithm for girls with adnexal masses.

CONTACTS AND LOCATIONS:
Overall Officials: KAREN NG, PI, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Takayasu H, Masumoto K, Tanaka N, Aiyoshi T, Sasaki T, Ono K, Chiba F, Urita Y, Shinkai T. A clinical review of ovarian tumors in children and adolescents. Pediatr Surg Int. 2020 Jun;36(6):701-709. doi: 10.1007/s00383-020-04660-w. Epub 2020 Apr 28. PMID 32346848
- [Background] Akakpo PK, Derkyi-Kwarteng L, Quayson SE, Gyasi RK, Anim JT. Ovarian Tumors in Children and Adolescents: A 10-Yr Histopathologic Review in Korle-Bu Teaching Hospital, Ghana. Int J Gynecol Pathol. 2016 Jul;35(4):333-6. doi: 10.1097/PGP.0000000000000257. PMID 26630227
- [Background] Amor F, Vaccaro H, Alcazar JL, Leon M, Craig JM, Martinez J. Gynecologic imaging reporting and data system: a new proposal for classifying adnexal masses on the basis of sonographic findings. J Ultrasound Med. 2009 Mar;28(3):285-91. doi: 10.7863/jum.2009.28.3.285. PMID 19244063
- [Background] Andreotti RF, Timmerman D, Strachowski LM, Froyman W, Benacerraf BR, Bennett GL, Bourne T, Brown DL, Coleman BG, Frates MC, Goldstein SR, Hamper UM, Horrow MM, Hernanz-Schulman M, Reinhold C, Rose SL, Whitcomb BP, Wolfman WL, Glanc P. O-RADS US Risk Stratification and Management System: A Consensus Guideline from the ACR Ovarian-Adnexal Reporting and Data System Committee. Radiology. 2020 Jan;294(1):168-185. doi: 10.1148/radiol.2019191150. Epub 2019 Nov 5. PMID 31687921
- [Background] Stankovic ZB, Sedlecky K, Savic D, Lukac BJ, Mazibrada I, Perovic S. Ovarian Preservation from Tumors and Torsions in Girls: Prospective Diagnostic Study. J Pediatr Adolesc Gynecol. 2017 Jun;30(3):405-412. doi: 10.1016/j.jpag.2017.01.008. Epub 2017 Jan 27. PMID 28137453
- [Background] Timmerman D, Testa AC, Bourne T, Ameye L, Jurkovic D, Van Holsbeke C, Paladini D, Van Calster B, Vergote I, Van Huffel S, Valentin L. Simple ultrasound-based rules for the diagnosis of ovarian cancer. Ultrasound Obstet Gynecol. 2008 Jun;31(6):681-90. doi: 10.1002/uog.5365. PMID 18504770
- [Background] Aldrink JH, Gonzalez DO, Sales SP, Deans KJ, Besner GE, Hewitt GD. Using quality improvement methodology to improve ovarian salvage for benign ovarian masses. J Pediatr Surg. 2017 Oct 10:S0022-3468(17)30638-3. doi: 10.1016/j.jpedsurg.2017.10.016. Online ahead of print. PMID 29106919